CLINICAL TRIAL: NCT06777927
Title: Effects of Exergaming Training on Balance Among Hypertensive Patients
Brief Title: Exergaming Training Among Hypertensive Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIPHAH/RCRS/REC/Letter-01198
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Hypertension
Keywords: Balance; Exergaming; Gait; Brain derived neurotrophic factor biomarker; Biopsychosocial
MeSH Terms: conditions — Hypertension | interventions — Exercise; Exergaming; Exercise Test

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): The group will not be provided with any interventions and would be used as controls.
  Interventions: Other: No intervention
- Conventional Exercise Training (Active Comparator): The subjects in the group would be doing treadmill training 3 days a week for 8 weeks (24 sessions) within target heart rate of moderate intensity.
  Interventions: Other: Exercise
- Exergaming Training Group (Experimental): The group would be doing exergaming 3 days a week for 8 weeks (24 sessions) within target heart rate of moderate intensity.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The participants would be playing exergames using XBOX-360 Kinect. Multiple games would be selected for the participants to play. The player would be upgraded to next levels of games after completing the initial levels.
  Other Names: Exergaming
  Arms: Exergaming Training Group
Other: Exercise — The subjects would be doing treadmill training within moderate intensity target heart rate.
  Other Names: Treadmill
  Arms: Conventional Exercise Training
Other: No intervention — The subjects would not be given any intervention and would be used as controls.
  Arms: Control group

SUMMARY:
Since Hypertension affects all body systems and importantly postural balance control. So, the evidence indicates a strong link and connection between balance and hypertension through somatosensory, visual, vestibular, musculoskeletal, and CNS integration of inputs from both peripheral and motor systems. Therefore, to fill this gap of how much balance and each of its aspects/components are affected, this study will be done for a detailed examination of this genuine integration and clinical interaction among hypertensive with game-based techniques on all three balance components (concerning Intensity, frequency, duration and dosage of VRET). Secondly, on the other hand (CR) programs, have shown very low compliance with recommended Physical Activity, which is why; by utilising this alternative, Virtual reality exergaming can be used as a quick, appropriate and equivalent alternative to traditional exercise programs. Also, in future, it could be suggested with promising effects in the provision of engaging, goal-oriented training for patients with hypertensive besides a sound, economical and clinically beneficial alternative to traditional Cardiac Rehabilitation. Finally, by exploring detailed clinical integration of Postural Balance with Hypertension using Virtual Reality the study will be able to highlight hypertension as a potent risk factor for future impaired balance and risks of falls. Thereby, hypertension's early identification (considering all biological, psychological, and social factors) and prevention may avert hypertensive to future debilitating complications and outcomes as a result of it.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Community dwelling controlled Hypertensive (particularly Stage 1, 130 to 139 (systolic) or 80 to 89 (diastolic) or Stage 2 hypertension from 140 or higher (systolic) or 90 (diastolic) if present with any (controlled diabetes or overweight patients) with a medical referral form for medical specialist with physiotherapeutic treatment provided by the local public or private healthcare system
2. Any race or gender with age 20 or older
3. No history of any orthopedic, neurological, Pulmonary or psychological disorders, Cognitive impairments etc.
4. Had not performed physical activity in the previous three months.

Exclusion criteria:

1. Grade III or grade IV heart failure according to the New York Heart Association (NYHA) Functional Classification.
2. Recent acute myocardial infarction; unstable angina; acute pericarditis. pulmonary hypertension; uncontrolled diabetes mellitus; Hypertensive crises or uncontrolled Hypertension or Pregnancy
3. Patients who had three consecutive absences during the intervention
4. Unable to answer or understand the gaming or exercise protocols and quality of life questionnaires and fulfil the exercise protocols, due to any severe cognitive deficit
5. Pain with ambulation or dizziness when standing or walking.
6. Contraindications to treadmill walking or VR gaming

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-10-16 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Gait and Balance App | Baseline before provision of interventions
  A new smartphone app (the Gait & Balance app) uses a structured and efficient protocol to evaluate performance during static balance and dynamic gait tasks that are commonly used in clinical practice. With the use of sensors embedded in standard smartphones, this technology has the potential to provide clinicians and sports professionals with easy access to more accurate and sensitive measures of balance and gait. This enhanced ability to assess and monitor progress may facilitate clinical decision making and optimize rehabilitation.
Gait and Balance App | After 4 weeks of interventions
  A new smartphone app (the Gait & Balance app) uses a structured and efficient protocol to evaluate performance during static balance and dynamic gait tasks that are commonly used in clinical practice. With the use of sensors embedded in standard smartphones, this technology has the potential to provide clinicians and sports professionals with easy access to more accurate and sensitive measures of balance and gait. This enhanced ability to assess and monitor progress may facilitate clinical decision making and optimize rehabilitation.
Gait and Balance App | After 8 weeks of interventions
  A new smartphone app (the Gait & Balance app) uses a structured and efficient protocol to evaluate performance during static balance and dynamic gait tasks that are commonly used in clinical practice. With the use of sensors embedded in standard smartphones, this technology has the potential to provide clinicians and sports professionals with easy access to more accurate and sensitive measures of balance and gait. This enhanced ability to assess and monitor progress may facilitate clinical decision making and optimize rehabilitation.
Brain-derived neurotrophic factor (BDNF) biomarker: | Baseline before provision of interventions
  Brain-Derived Neurotrophic Factor (BDNF) is a protein of the neurotrophin family encoded by the BDNF gene that plays an important role in the modulation of synaptic plasticity processes underlying learning, memory, and behavior. This protein plays a fundamental role in neurodevelopment, acting on neurogenesis and on the differentiation and maturation of neurotransmitter systems such as the brain stress system and the brain reward and motivation system. Evidence shows that BDNF reduced levels are linked to reduced synaptic plasticity and neuronal atrophy, while elevated levels are associated with survival and neuronal differentiation and brain plasticity.
Brain Derived Neurotrophic Factor Biomarker | After 8 weeks of interventions
  Brain-Derived Neurotrophic Factor (BDNF) is a protein of the neurotrophin family encoded by the BDNF gene that plays an important role in the modulation of synaptic plasticity processes underlying learning, memory, and behavior. This protein plays a fundamental role in neurodevelopment, acting on neurogenesis and on the differentiation and maturation of neurotransmitter systems such as the brain stress system and the brain reward and motivation system. Evidence shows that BDNF reduced levels are linked to reduced synaptic plasticity and neuronal atrophy, while elevated levels are associated with survival and neuronal differentiation and brain plasticity.
Exercise Enjoyment Questionnaire (EEQ) | After 8 weeks of interventions
  Exergame Enjoyment Questionnaire (EEQ), a new 20-item questionnaire for measuring how much players enjoyed an exergame. Thus, the minimum score is 20 points, and the maximum score is 100 points. Higher is better, indicating more enjoyment. Questions are intended to be administered to users immediately after playing an exergame with a high average agreement percentage per question (of ~85%), EEQ will only be taken in Exergaming Group after 8 weeks of intervention.
The Montreal Cognitive Assessment (MoCA) | Baseline before provision of interventions
  It is a validated brief cognitive screening measure that is commonly employed in clinical practice and research settings. The MoCA evaluates several cognitive domains including visuospatial ability, executive functioning, language, memory, attention, and orientation. 18-25 points: Mild cognitive impairment. 10-17 points: Moderate cognitive impairment. Fewer than 10 points: Severe cognitive impairment.
Montreal Cognitive Assessment (MoCA) | After 4 weeks of interventions
  It is a validated brief cognitive screening measure that is commonly employed in clinical practice and research settings. The MoCA evaluates several cognitive domains including visuospatial ability, executive functioning, language, memory, attention, and orientation. 18-25 points: Mild cognitive impairment. 10-17 points: Moderate cognitive impairment. Fewer than 10 points: Severe cognitive impairment.
Montreal Cognitive Assessment (MoCA) | After 8 weeks of interventions
  It is a validated brief cognitive screening measure that is commonly employed in clinical practice and research settings. The MoCA evaluates several cognitive domains including visuospatial ability, executive functioning, language, memory, attention, and orientation. 18-25 points: Mild cognitive impairment. 10-17 points: Moderate cognitive impairment. Fewer than 10 points: Severe cognitive impairment.
3 Min Walk Test | Baseline before provision of interventions
  The three-minute walk test has proven to be reproducible and is well tolerated by patients. It evaluates the distance a person can walk on a flat, rigid surface in 3 minutes. Its main objective is to determine exercise tolerance and oxygen saturation during submaximal exercise
3 Min Walk Test | After 4 weeks of interventions
  The three-minute walk test has proven to be reproducible and is well tolerated by patients. It evaluates the distance a person can walk on a flat, rigid surface in 3 minutes. Its main objective is to determine exercise tolerance and oxygen saturation during submaximal exercise
3-min walk Test | After 8 weeks of interventions
  The three-minute walk test has proven to be reproducible and is well tolerated by patients. It evaluates the distance a person can walk on a flat, rigid surface in 3 minutes. Its main objective is to determine exercise tolerance and oxygen saturation during submaximal exercise
Social Functioning Questionnaire (SFQ) | Baseline before provision of interventions
  Inventory/Questionnaire, each of the 8 items of the SFQ is scored on a four- point scale (0-3) with a total possible score of 24. The Social Functioning is a Rapid and Robust Measure of Perceived Functioning. Test content may be reproduced and used for non-commercial research and educational purposes without seeking written permission. Distribution must be controlled, meaning only to the participants engaged in the research or enrolled in the educational activity. The Social Functioning Questionnaire (SFQ), an eight-item self-report scale (score range 0-24), is a semi- structured interview which has been used primarily with non-psychotic patients and has good test-retest and inter-rater reliability as well as construct validity. It is a quick assessment of perceived social function.
Social Functioning Questionnaire (SFQ) | After 4 weeks of interventions
  Inventory/Questionnaire, each of the 8 items of the SFQ is scored on a four- point scale (0-3) with a total possible score of 24. The Social Functioning is a Rapid and Robust Measure of Perceived Functioning. Test content may be reproduced and used for non-commercial research and educational purposes without seeking written permission. Distribution must be controlled, meaning only to the participants engaged in the research or enrolled in the educational activity. The Social Functioning Questionnaire (SFQ), an eight-item self-report scale (score range 0-24), is a semi- structured interview which has been used primarily with non-psychotic patients and has good test-retest and inter-rater reliability as well as construct validity. It is a quick assessment of perceived social function.
Social Functioning Questionnaire (SFQ) | After 8 weeks of interventions
  Inventory/Questionnaire, each of the 8 items of the SFQ is scored on a four- point scale (0-3) with a total possible score of 24. The Social Functioning is a Rapid and Robust Measure of Perceived Functioning. Test content may be reproduced and used for non-commercial research and educational purposes without seeking written permission. Distribution must be controlled, meaning only to the participants engaged in the research or enrolled in the educational activity. The Social Functioning Questionnaire (SFQ), an eight-item self-report scale (score range 0-24), is a semi- structured interview which has been used primarily with non-psychotic patients and has good test-retest and inter-rater reliability as well as construct validity. It is a quick assessment of perceived social function.
SF -36 Quality of Life Questionnaire | Baseline before provision of interventions
  The SF-36 is a self-reported outcome measure assessing the impact of health on an individual everyday life. It is often used as a quality-of-life measure. The SF- 36 uses eight domains: used as a general measure of health so can be used with the general population. It is a promising instrument for measuring health perception in a general population. It is easy to use, acceptable to patients, and fulfils stringent criteria of reliability and validity. To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
SF -36 Quality of Life Questionnaire | After 4 weeks of interventions
  The SF-36 is a self-reported outcome measure assessing the impact of health on an individual everyday life. It is often used as a quality-of-life measure. The SF- 36 uses eight domains: used as a general measure of health so can be used with the general population. It is a promising instrument for measuring health perception in a general population. It is easy to use, acceptable to patients, and fulfils stringent criteria of reliability and validity. To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
SF -36 Quality of Life Questionnaire | After 8 weeks of interventions
  The SF-36 is a self-reported outcome measure assessing the impact of health on an individual everyday life. It is often used as a quality-of-life measure. The SF- 36 uses eight domains: used as a general measure of health so can be used with the general population. It is a promising instrument for measuring health perception in a general population. It is easy to use, acceptable to patients, and fulfils stringent criteria of reliability and validity. To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
Timed up and Go (TUG) | Baseline before provision of interventions
  This test measures the dynamic balance and functional mobility in older adults, as well as in the neurological population. The Timed Up & Go Test has been found to be correlated with falls and those who require 30 s or more to complete the Timed Up & Go tend to be dependent on others for care
Timed up and Go (TUG) | After 4 weeks of interventions
  This test measures the dynamic balance and functional mobility in older adults, as well as in the neurological population. The Timed Up & Go Test has been found to be correlated with falls and those who require 30 s or more to complete the Timed Up & Go tend to be dependent on others for care
Timed up and Go (TUG) | After 8 weeks of interventions
  This test measures the dynamic balance and functional mobility in older adults, as well as in the neurological population. The Timed Up & Go Test has been found to be correlated with falls and those who require 30 s or more to complete the Timed Up & Go tend to be dependent on others for care
Berg Balance Scale (BBS) | Baseline before provision of interventions
  The Berg balance scale helps determine one's ability to balance safely. The Berg balance scale was created in 1989, it was intended to assess both balance and fall risk. The scale consists of 14 tasks that a healthcare provider scores on a scale from 0 to 4. The higher the score, the better is the better is the balance. The highest possible score is 56. The Berg balance scale test takes about 15 to 20 minutes to complete. 0 to 20: A person with a score in this range will likely need the assistance of a wheelchair to move around safely. 21 to 40: A person with a score in this range will need some type of walking assistance, like a cane or a walker. 41 to 56: A person with a score in this range is considered independent and should be able to move around safely without assistance. It is widely used in clinical settings and is much valid and reliable.
Berg Balance Scale (BBS) | After 4 weeks of interventions
  The Berg balance scale helps determine one's ability to balance safely. The Berg balance scale was created in 1989, it was intended to assess both balance and fall risk. The scale consists of 14 tasks that a healthcare provider scores on a scale from 0 to 4. The higher the score, the better is the better is the balance. The highest possible score is 56. The Berg balance scale test takes about 15 to 20 minutes to complete. 0 to 20: A person with a score in this range will likely need the assistance of a wheelchair to move around safely. 21 to 40: A person with a score in this range will need some type of walking assistance, like a cane or a walker. 41 to 56: A person with a score in this range is considered independent and should be able to move around safely without assistance. It is widely used in clinical settings and is much valid and reliable.
Berg Balance Scale (BBS) | After 8 weeks of interventions
  The Berg balance scale helps determine one's ability to balance safely. The Berg balance scale was created in 1989, it was intended to assess both balance and fall risk. The scale consists of 14 tasks that a healthcare provider scores on a scale from 0 to 4. The higher the score, the better is the better is the balance. The highest possible score is 56. The Berg balance scale test takes about 15 to 20 minutes to complete. 0 to 20: A person with a score in this range will likely need the assistance of a wheelchair to move around safely. 21 to 40: A person with a score in this range will need some type of walking assistance, like a cane or a walker. 41 to 56: A person with a score in this range is considered independent and should be able to move around safely without assistance. It is widely used in clinical settings and is much valid and reliable.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Foundation University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No